CLINICAL TRIAL: NCT06030505
Title: Effectiveness of Nirsevimab in Children Hospitalised With RSV Bronchiolitis
Acronym: ENVIE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: ENVIE; 2023-A01803-42 (Other: ID-RCB)
Record Dates: First submitted 2023-08-24; First posted 2023-09-11 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2024-04

CONDITIONS: Bronchiolitis, Viral
MeSH Terms: conditions — Bronchiolitis, Viral

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case patients: Collection of medical data in a non-identifying way (demographic data, medical history, clinical data, microbiological data) to meet the objectives of the research.
  Interventions: Other: No intervention required by the protocol
- Control patients: Collection of medical data in a non-identifying way (demographic data, medical history, clinical data, microbiological data) to meet the objectives of the research.
  Interventions: Other: No intervention required by the protocol

INTERVENTIONS:
Other: No intervention required by the protocol — No visits or samples will be taken specifically for this study. This research involves only prospective or retrospective data collection in relation to the usual hospital management of the child included. Similarly, patient follow-up will be strictly within the framework of their usual hospital care in relation to their pathology.

SUMMARY:
Respiratory tract infections caused by respiratory syncytial virus (RSV) are a worldwide burden and represent a major public health issue. In France, bronchiolitis is responsible for around 100,000 emergency room visits and 50,000 hospital admissions every year; 75% of infants hospitalised for RSV bronchiolitis are healthy full-term children.

Recent discoveries concerning the specific viral epitopes of RSV have made it possible to move from an empirical approach to a targeted preventive or curative approach (monoclonal antibodies, vaccines, anti-viral drugs).

Nirsevimab is a monoclonal antibody against RSV with enhanced neutralising activity and a prolonged half-life. A randomised, placebo-controlled phase III trial demonstrated the effectiveness of nirsevimab in reducing lower respiratory tract infections caused by RSV requiring medical management in healthy premature and term infants, with a favourable safety profile. The US Food and Drug Administration (FDA) approved the first RSV vaccine on May 3, 2023, and the second was approved on May 31, 2023. Nirsevimab was approved by the European Medicines Agency (EMA) on November 4, 2022.

ELIGIBILITY:
Inclusion Criteria:

Cases :

* Children under 12 months of age
* Treated for acute RSV bronchiolitis
* Hospitalised following a visit to the paediatric emergency department

Controls :

* Children under 12 months
* Hospitalised in the conventional sector or in a short-stay hospital unit, or having consulted a paediatric emergency department for one of the following reasons
* Febrile urinary tract infection, without acute ear, nose, and throat (ENT) or respiratory symptoms
* Acute gastroenteritis, without acute ENT or respiratory symptoms
* Infant colic without fever, without ENT or acute respiratory symptoms
* Stagnant weight or feeding difficulties without fever, acute ENT or respiratory symptoms
* Neonatal jaundice without fever or acute ENT or respiratory symptoms
* Unexplained crying without fever, without ENT or acute respiratory symptoms
* Head injury, without acute ENT or respiratory symptoms
* Patient hospitalised for acute surgery without fever, without ENT or acute respiratory symptoms

Exclusion Criteria:

* Refusal to participate by the patient, their relative or legal representative
* Administration of Palivizumab.
* Maternal vaccination against RSV.

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Paediatric patients under 12 months of age treated for RSV bronchiolitis (for cases), or for one of the conditions listed in the inclusion criteria (for controls).
Sampling Method: Non-Probability Sample
Enrollment: 1140 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Proportion of patients passively immunised with nirsevimab | 7 days
  Proportion of patients passively immunised with nirsevimab in children hospitalised with RSV bronchiolitis and in the control group

SECONDARY OUTCOMES:
Proportion of hospitalised children for RSV bronchiolitis requiring invasive or non-invasive ventilatory passively immunised with nirsevimab | 7 days
  Proportion of children passively immunised with nirsevimab hospitalised for bronchiolitis requiring invasive or non-invasive ventilatory support, including RSV bronchiolitis
Length of hospital stay | 7 days
  Length of hospital stay for children with RSV bronchiolitis.
Time immunisation | 7 days
  Time between immunisation with nirsevimab and hospitalisation for RSV bronchiolitis.
Frequency of hospital admissions | 7 days
  Monthly frequency of hospital admissions for RSV bronchiolitis among participating centres over time
Proportion of children hospitalised for RSV bronchiolitis with viral co-detection | 7 days
  Proportion of children hospitalised for RSV bronchiolitis with viral co-detection or viral detection other than RSV on nasopharyngeal swab

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - CHU Bondy - Jean Verdier, Bondy
  - CHI Créteil, Créteil
  - Hôpital Armand Trousseau AP-HP, Paris
  - CHU Robert-Debré, Paris
  - CHU Toulouse-hôpital des Enfants, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Assad Z, Romain AS, Aupiais C, Shum M, Schrimpf C, Lorrot M, Corvol H, Prevost B, Ferrandiz C, Giolito A, Valtuille Z, Bendavid M, Cohen JF, Toubiana J, de Pontual L, Delande CF, Levy M, See P, Cohen R, Levy C, Angoulvant F, Lenglart L, Gits-Muselli M, Biran V, Diallo K, Alemede O, El Hebil MM, Durrmeyer X, Labouret G, Casanovas N, Hallak B, Marechal O, Jung C, Brehin C, Ouldali N. Nirsevimab and Hospitalization for RSV Bronchiolitis. N Engl J Med. 2024 Jul 11;391(2):144-154. doi: 10.1056/NEJMoa2314885. PMID 38986058